CLINICAL TRIAL: NCT04371471
Title: On-admission Multifactorial Evaluation of Inflammation as Prognostic Marker of Death in Patients Diagnosed With Coronavirus Infectious Disease (COVID-19) Syndrome
Brief Title: Pandemic Triage Score in Patients With Known or Suspected Severe Acute Respiratory Syndrome (SARS) CoronaVirus (CoV) 2 Infection
Acronym: STC-19
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier de la Rochelle Ré Aunis (Other)
Collaborators: NumaHealth International (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020/P04/288
Record Dates: First submitted 2020-04-30; First posted 2020-05-01 (Actual); Results first posted 2022-04-07 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: SARS-CoV-2 Acute Respiratory Disease; Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with COVID-19: Patient with clinical signs of CoV-2-SARS infection and signs of severity
  Interventions: Diagnostic Test: STC-19 score

INTERVENTIONS:
Diagnostic Test: STC-19 score — Score calculated by an algorithm using a vital sign (systolic blood pressure) and biomarkers (complete blood count with differential)

SUMMARY:
During this pandemic period, the goal of the health care system is to optimize the use of intensive care services for patients infected with SARS-CoV-2, given the frequency of complications that can lead to high mortality.

When patients with suspected or confirmed COVID-19 are admitted to hospital, whether or not they are symptomatic, there is currently no method to predict who will progress to complications requiring the use of intensive measures in 24-48 hours.

DETAILED DESCRIPTION:
The body undergoes a systemic adaptation response to severe illness. Elevated cortisol and systemic inflammation are two key responses. Along with hypotension, this triad can lead to end-organ failure and death in critical illness. In critical illness, serum cortisol is dissociated from its tissular activity. We have developed a formula that calculates tissular action of cortisol called the cortisol index. It correlates in chronic ambulatory illness, and acute illness such as myocardial infarction (manuscript pending). Elevated neutrophil to lymphocyte ration (NLR) is a marker of systemic inflammation and predictor of mortality on admission to the emergency department. We have confirmed this in a retrospective and prospective study (manuscript pending, data available upon request).

The purpose of this study is to evaluate a triage score (STC-19) based on patients' biological state at the time of diagnosis, to objectively determine which patients are most likely to require intensive medical services within 24-48 hours of presentation of the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Patient with clinical signs of CoV-2-SARS infection
* Complete blood count test and systolic blood pressure available at the time of diagnosis
* Informed of the study.

Exclusion Criteria:

* Women beyond the 1st trimester of pregnancy
* Persons under-the-age-of or legally-denied medical decision-making capacity by a judicial or administrative decision,
* Persons of full age who are subject to a legal protection measure,
* Persons unable to consent,
* Persons who are not members of or beneficiaries of a social welfare program administered by the Republic of France
* Patient's refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with clinical signs of CoV-2-SARS infection and signs of severity (polypnea, saturation < 90% room air, dyspnea, systolic blood pressure < 90 mmHg, altered consciousness, somnolence, confusion) and/or co-morbidities (> 70 years of age, Respiratory pathology at risk of decompensation, Chronic renal failure on dialysis, Heart failure or IV, Cirrhosis ≥ B, Cardiovascular history, Diabetes with poor balance or co-morbidities, Immunosuppression, Dementia)
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Chalvet, MD, Study Director — Numa Health International; Kamyar M. Hedayat, MD, Study Director — Numa Health International; Jean-Claude Lapraz, MD, Study Director — Numa Health International; Serge Bénéteaud, MD, Principal Investigator — Groupe Hospitalier de la Rochelle Ré Aunis
Locations (1):
- Groupe Hospitalier de la Rochelle Ré Aunis, La Rochelle, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available with publication. A Digital Object Identifier will be used. Keyword are SARS-Cov2, COVID-19, cortisol, systemic inflammation, hypotension, complete blood count.
  The only available version will be the locked database. With the exception of dates, all data will be made available. Dates will only be collected to verify the quality of the clinical trial execution. They do not add to the clinical question, and may be a means of indirectly identifying patients.
  The database will be made available through a secure cloud-based repository (Mendeley Data) which is an open research data repository accessible online, where researchers can upload and share their research data.
  Medical Subject Headings (MESH) terms will be used to describe clinical data. Methodology for calculating the STC-19 score will be provided in the publication.
  International standard unit will be used.
Supporting Information: CSR
Time Frame: Data will be made available with publication and up to 15 years after the end of the study
Access Criteria: A Digital Object Identifier will be provided

REFERENCES:
- [Background] Selye H. THE SIGNIFICANCE OF THE ADRENALS FOR ADAPTATION. Science. 1937 Mar 5;85(2201):247-8. doi: 10.1126/science.85.2201.247. No abstract available. PMID 17841381
- [Background] Peeters B, Langouche L, Van den Berghe G. Adrenocortical Stress Response during the Course of Critical Illness. Compr Physiol. 2017 Dec 12;8(1):283-298. doi: 10.1002/cphy.c170022. PMID 29357129
- [Background] Oakley RH, Cidlowski JA. The biology of the glucocorticoid receptor: new signaling mechanisms in health and disease. J Allergy Clin Immunol. 2013 Nov;132(5):1033-44. doi: 10.1016/j.jaci.2013.09.007. Epub 2013 Sep 29. PMID 24084075
- [Background] Groeneweg FL, Karst H, de Kloet ER, Joels M. Rapid non-genomic effects of corticosteroids and their role in the central stress response. J Endocrinol. 2011 May;209(2):153-67. doi: 10.1530/JOE-10-0472. Epub 2011 Feb 28. PMID 21357682
- [Background] de Jager CP, van Wijk PT, Mathoera RB, de Jongh-Leuvenink J, van der Poll T, Wever PC. Lymphocytopenia and neutrophil-lymphocyte count ratio predict bacteremia better than conventional infection markers in an emergency care unit. Crit Care. 2010;14(5):R192. doi: 10.1186/cc9309. Epub 2010 Oct 29. PMID 21034463
- [Background] de Jager CP, Wever PC, Gemen EF, Kusters R, van Gageldonk-Lafeber AB, van der Poll T, Laheij RJ. The neutrophil-lymphocyte count ratio in patients with community-acquired pneumonia. PLoS One. 2012;7(10):e46561. doi: 10.1371/journal.pone.0046561. Epub 2012 Oct 1. PMID 23049706
- [Result] Hedayat KM, Chalvet D, Yang M, Golshan S, Allix-Beguec C, Beneteaud S, Schmit T. Evolution of Modeled Cortisol Is Prognostic of Death in Hospitalized Patients With COVID-19 Syndrome. Front Med (Lausanne). 2022 Jun 6;9:912678. doi: 10.3389/fmed.2022.912678. eCollection 2022. PMID 35733873

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient With Covid-19
Started | 91
Completed | 81
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | Patient With Covid-19
Number analyzed (Participants) | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 59
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 91
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27.2 (5.4)
Hypertension [Count of Participants; unit: Participants] | 54
Diabetes [Count of Participants; unit: Participants] | 67
Chronic respiratory disease [Count of Participants; unit: Participants] | 71

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Normal and Above Triage (STC-19) Score
Description: Correlation between the STC-19 score based on biological measures at the time of diagnosis and patient outcome (deceased or alive within 29 days of hospitalization)
  The STC-19 score is based on the genito-thyroid index (GTi) calculated from the neutrophil-to-lymphocyte ratio (NLR) and the cortisol index :
  Normal value for cortisol range from 3 to 7 Normal value for GTi range from 1.5 to 2.5
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Groups:
- Alive Within 29 Days of Hospitalization: Patients admitted through the emergency department and confirmed to be positive for SARS CoV-2.
  Still living at day 29 after hospitalization
- Death Within 29 Days of Hospitalization: Patients admitted through the emergency department and confirmed to be positive for SARS CoV-2.
  Death due to coronavirus disease (COVID-19) was defined as death prior to day 29.
  Any deaths from day 29 days onward were considered as death from complications of COVID-19.
Arm/Group | Alive Within 29 Days of Hospitalization | Death Within 29 Days of Hospitalization
Number analyzed (Participants) | 56 | 25
Participants
  Genito-thyroid index: Normal value | 52 | 12
  Genito-thyroid index: Above normal value | 4 | 5
  Genito-thyroid index: Missing data | 0 | 8
  Cortisol index adjusted: Normal value | 55 | 0
  Cortisol index adjusted: Above normal value | 0 | 21
  Cortisol index adjusted: Missing data | 1 | 4

2. Secondary Outcome: Number of Participants With Normal and Above Genito-thyroid Index (GTi) Value
Description: Correlation between the STC-19 score based on biological measures at the time of diagnosis and patient outcome (deceased or alive within 29 days of hospitalization) The genito-thyroid index (GTi) is calculated from the neutrophil-to-lymphocyte ratio (NLR).
  Normal value for GTi range from 1.5 to 2.5
Time Frame: Day 5
Measure: Count of Participants; unit: Participants
Groups:
- Death Within 29 Days of Hospitalization: Patients admitted through the emergency department and confirmed to be positive for SARS CoV-2.
  Death due to COVID-19 was defined as death prior to day 29. Any deaths from day 29 days onward were considered as death from complications of COVID-19.
Arm/Group | Alive Within 29 Days of Hospitalization | Death Within 29 Days of Hospitalization
Number analyzed (Participants) | 56 | 25
Participants
  Normal value | 33 | 4
  Above normal value | 11 | 10
  Missing data | 12 | 11

ADVERSE EVENTS:
Time Frame: 28 days
Groups:
- Patient With Covid-19: Patient with clinical signs of CoV-2-SARS infection and signs of severity
  STC-19 score: Score calculated by an algorithm using biomarkers
Arm/Group | Patient With Covid-19
All-Cause Mortality (participants affected / at risk) | 25/81
Serious Adverse Events (participants affected / at risk) | 0/81
Other Adverse Events (participants affected / at risk) | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT04371471/Prot_SAP_000.pdf